CLINICAL TRIAL: NCT06460571
Title: The Effect of Cardiac Rehabilitation With and Without Delorme Technique of Progressive Resisted Exercises to Improve Dyspnea and Quality of Life in Patients of Post PCI.
Brief Title: Cardiac Rehabilitation With and Without Delorme Technique of Progressive Resisted Exercises in Patients of Post PCI.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0365
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Percutaneous CORONARY INTERVENTION
Keywords: Quality of Life; Cardiac Rehabilitation; Delorme Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Cardiac rehabilitation with Delorme technique (Experimental): The intervention group will receive Delorme technique along with standard cardiac rehabilitation, involving 10 repetition max of aerobic exercises, resistance exercises of 10 minutes will be given in each training session
  Interventions: Other: Standard Cardiac rehabilitation with Delorme technique; Other: standard cardiac rehabilitation
- standard cardiac rehabilitation (Active Comparator): The control group (Group B) will undergo standard cardiac rehabilitation (outpatient cardiac rehabilitation) which include walking, cycling and strength training which will have 5-10 minutes warm-up followed by training for 30-45 minutes, concluding with cool-down without the Delorme technique.
  Interventions: Other: standard cardiac rehabilitation

INTERVENTIONS:
Other: Standard Cardiac rehabilitation with Delorme technique — Aerobic training will be provided three alternate days a week at 60-70% of maximum heart rate for eight weeks. Resistance training for 3 sets and 10 repetitions (10 lifts with 50%of 10RM, then 75% of 10RM and will progress to 100% of 10RM) will involve seven exercises (abdominal curl ups, bicep curls, triceps extension, back extension, leg curls, side leg raises and knee extensions).
  Arms: Standard Cardiac rehabilitation with Delorme technique
Other: standard cardiac rehabilitation — The control group (Group B) will undergo standard cardiac rehabilitation (outpatient cardiac rehabilitation) which include walking, cycling and strength training which will have 5-10 minutes warm-up followed by training for 30-45 minutes, concluding with cool-down without the Delorme technique. The control group will not perform any specific training but will be given a diet chart to follow

SUMMARY:
To find the effect of cardiac rehabilitation program with and without progressive resisted exercises on patients after acute stage of PCI with at least 8 weeks history. It is a randomized clinical trial using convenient sampling technique. Randomly assign participants into two groups: An intervention group receiving Delorme progressive resisted exercise along with cardiac rehab and a control group undergoing standard cardiac rehabilitation alone. In Group A, Delorme technique will involve a 10-repetition max of aerobic and resistance exercises along with cardiac rehab. Seven different exercises will be performed in 3 sets of 10-repetition max. The control group will not be performing any type of training but will undergo cardiac rehab alone. Data will be analyzed using t test and SPSS 21 will be used for data collection. Age group will be from ≥70 years with patient undergoing dyspnea along with recent history of primary diseases. Data will be collected from Bethania Hospital, Sialkot through tools like the 6-minute walk test, Rose Angina questionnaire or settle angina questionnaire, quality of life scale (QOLFS), and Modified Borg dyspnea scale.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 70 years"
* "Recent history of PCI due to primary diseases (coronary heart disease, acute myocardial infarction, acute coronary syndrome, acute angina)"
* "Presence of dyspnea"
* "First-time PCI

Exclusion Criteria:

* "Renal failure"
* Chronic liver disease
* Chest disease
* Patient who could not fulfill the questionnaire or cooperate through the performed procedures

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
QUALITY OF LIFE SCALE: | baseline and fourth week
  "The QOLS was originally a 15-item instrument that measured five conceptual domains of quality of life: material and physical well-being, relationships with other people, social, community and civic activities, personal development and fulfillment, and recreation
MODIFIED BORG DYSPNEA SCALE | baseline and fourth week
  The Modified Borg Dyspnea Scale (MBS) is a numerical rating system (0-10) assessing dyspnea during submaximal exercise. Administered with the six-minute walk test (6MWT), a common measure for pulmonary arterial hypertension (PAH), the MBS is consistent within a single session
SETTLE ANGINA QUESTIONNAIRE | baseline and fourth week
  Settle Angina Questionnaire (SAQ) scale is a disease specific scale is a diabetes specific scale for assessing QOL of CHD patients; have 5 items covering domains; Physical Limitation, Angina Stability, Angina Severity, Treatment Satisfaction and Disease Perception

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Bethania Hospital,, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fish DE, Krabak BJ, Johnson-Greene D, DeLateur BJ. Optimal resistance training: comparison of DeLorme with Oxford techniques. Am J Phys Med Rehabil. 2003 Dec;82(12):903-9. doi: 10.1097/01.PHM.0000098505.57264.DB. PMID 14627926
- [Background] Jelinek HF, Huang ZQ, Khandoker AH, Chang D, Kiat H. Cardiac rehabilitation outcomes following a 6-week program of PCI and CABG Patients. Front Physiol. 2013 Oct 30;4:302. doi: 10.3389/fphys.2013.00302. eCollection 2013. PMID 24198786